CLINICAL TRIAL: NCT05507749
Title: Cyroablation for Pulmonary Vein Isolation Alone in Patients with Early Persistent AF Assessed by Continuous Monitoring
Acronym: COOL-PER
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: Seoul National University Bundang Hospital (Other); Samsung Medical Center (Other); Hallym University Medical Center (Other); Asan Medical Center (Other)
Responsible Party: Principal Investigator, Eue-Keun Choi, Professor, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: COOL PER
Record Dates: First submitted 2022-08-08; First posted 2022-08-19 (Actual); Last update posted 2024-11-06 (Actual); Status verified 2024-11

CONDITIONS: Atrial Fibrillation, Persistent
Keywords: Cryoablation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- a group of participants receive implantable loop recorder before cryoballoon ablation (Experimental): Following enrollment, an implantable loop recorder is implanted in all participants for the purpose of arrhythmia (any atrial fibrillation or atrial tachycardia) detection (Reveal LINQ, Medtronic, Minneapolis, MN).
  Interventions: Procedure: cryoballoon ablation; Device: implantable loop recorder insertion

INTERVENTIONS:
Procedure: cryoballoon ablation — Cryoballoon ablation for the treatment of atrial fibrillation
Device: implantable loop recorder insertion — The device called a implantable loop recorder, is placed just under the skin of one's chest during a minor surgery.

SUMMARY:
This study aimed to evaluate the efficacy of Cryoablation in patients with early persistent atrial fibrillation as a first index procedure using continuous cardiac rhythm monitoring.

DETAILED DESCRIPTION:
Atrial fibrillation is the most common cardiac arrhythmia. With the population aging, the prevalence of atrial fibrillation is increasing globally. Recently, Cryoablation has been demonstrated non-inferior efficacy and safety compared with catheter ablation in atrial fibrillation patients. Cryoablation with the simplicity of the procedure brought the substantial shortening of the total procedure time compared to catheter ablation with comparable long-term atrial fibrillation free survival and procedure-related adverse events. However, most of the previous studies that reported non-inferior efficacy and safety of Cryoablation versus catheter ablation were only included patients with paroxysmal atrial fibrillation. The long-term efficacy of Cryoablation in patients with persistent atrial fibrillation is controversial.

In patients with persistent atrial fibrillation, pulmonary vein isolation alone showed comparable atrial fibrillation recurrence rate compared to pulmonary vein isolation with additional ablation, including linear ablation or ablation of complex fractionated electrograms.

In a recent study, Cryoablation was safe and had good outcomes in patients with persistent and long-standing persistent atrial fibrillation within relatively short procedure time; atrial fibrillation recurrence rate was 36% in persistent atrial fibrillation and 43% in long-standing persistent atrial fibrillation. Among patients with persistent atrial fibrillation ≤1 year, pulmonary vein isolation using cryoballoon had 39% of any atrial fibrillation/atrial tachycardia recurrence rate during a 1-year follow-up. Pre-predictor such as smaller left atrium size or atrial fibrillation history less than three years was associated with a better outcome of atrial fibrillation cryoablation. Therefore, early ablation of persistent atrial fibrillation using Cryoablation may be related to a good outcome that is nearly comparable to those with paroxysmal atrial fibrillation. Namely, pulmonary vein isolation by Cryoablation could be reasonable as the first procedure in patients with early persistent atrial fibrillation. Based on the results of the STOP Persistent atrial fibrillation trial, the Arctic Front Advance cryoablation system (Medtronic) was granted an expanded indication by the US Food and Drug Administration for the treatment of recurrent, drug-refractory, symptomatic, persistent atrial fibrillation. It is the first ablation catheter in the United States to receive an indication for persistent-as opposed to paroxysmal-atrial fibrillation.

Not only atrial fibrillation recurrence merely defined as any atrial fibrillation episode lasting 30 seconds or more, but the atrial fibrillation burden is also a relevant indicator for evaluation of procedure success. Among patients with paroxysmal atrial fibrillation, a recent prospective study reported that atrial fibrillation burden dramatically decreased after Cryoablation by 99% . There was limited data about the efficacy of Cryoablation in patients with early persistent atrial fibrillation evaluated by actual atrial fibrillation burden using continuous cardiac rhythm monitoring.

ELIGIBILITY:
Inclusion Criteria:

* Drug refractory symptomatic persistent atrial fibrillation diagnosed within 3 years
* Either two conditions

  1. atrial fibrillation episode lasting longer than 7 days, but less than 3 years documented by consecutive electrocardiogram recordings of 100% atrial fibrillation greater than 7 days apart or
  2. atrial fibrillation episode requiring electrical or pharmacological cardioversion after 24 hours of atrial fibrillation documented by continuous recording
* Willing to comply with study requirements and give informed consent to participate in this clinical study

Exclusion Criteria:

* Long-standing persistent atrial fibrillation more than 3 years
* Sinus rhythm at enrollment
* Recurrent sinus rhythm after electrical cardioversion
* Severe left ventricular dysfuncion (left ventricle ejection fraction < 30%)
* Previous ablation procedure or surgery for atrial fibrillation
* Contraindication to chronic anticoagulation therapy or heparin
* Documented left atrial diameter >50 mm from parasternal long-axis view
* A percutaneous coronary intervention or myocardial infarction ≤3 months
* A stroke or transient ischemic attack ≤6 months
* Planned cardiovascular intervention
* Mental or physical inability to participate in the study
* Participation in another randomized clinical trial
* Uncontrolled hypertension, untreated hypothyroidism or hyperthyroidism
* Requirement for dialysis due to terminal renal failure

Ages: 20 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2020-11-27 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Change of implantable cardiac monitor-detected atrial fibrillation/atrial flutter burden. | After cryoablation (between 3-month and 1-year) and pre-ablation
  The percentage of time spent in atrial fibrillation (hours of atrial fibrillation/hours of monitoring) during the first year after pulmonary vein isolation (excluding a 3-month window) compared to pre-ablation atrial fibrillation/atrial flutter burden.

SECONDARY OUTCOMES:
Time to the first recurrence of atrial fibrillation/atrial flutter | From 3-month after cryoablation to the removal of the implantable loop recorder, up to 3years.
  Atrial fibrillation/atrial flutter recurrence, defined as an episode of atrial arrhythmia beyond the first 3 months post-ablation (blanking period), lasting for 30 seconds or more
Recurrence nature of atrial fibrillation | From 3-month after cryoablation to the removal of the implantable loop recorder, up to 3years.
  paroxysmal atrial fibrillation or persistent atrial fibrillation
36-Item Short Form Health Survey composite scores | Pre-ablation and 1-year after ablation
  Quality of life assessed with the use of the Medical Outcomes Study 36-Item Short-From Health Survey [SF-36]; range 0 to 100, with higher scores indicating better quality of life
European Heart Rhythm Association score | Pre-ablation and 1-year after ablation
  The European Heart Rhythm Association score of atrial fibrillation (or EHRA score) is a classification system for the extent of atrial fibrillation. It places patients in one of four categories based on how much they are limited during physical activity; the limitations/symptoms are in regard to normal breathing and varying degrees in shortness of breath and/or angina.
  EHRA Class / Symptoms I- No symptoms. II- Mild symptoms; normal daily activity not affected. III- Severe symptoms; normal daily activity affected. IV- Disabling symptoms; normal daily activity discontinued.
Atrial fibrillation/atrial flutter recurrence and changes in atrial fibrillation/atrial flutter burden | From 3-month after cryoablation to the removal of the implantable loop recorder, up to 3years.
  Atrial fibrillation/atrial flutter recurrence and changes in AF/AT burden from 3-month after cryoablation to the removal of the implantable loop recorder

CONTACTS AND LOCATIONS:
Overall Officials: Eue-Keun Choi, M.D. Ph.D., Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National university Hostpital, Seoul, Jongno-gu, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lee SR, Choi EK, Lee KY, Choi J, Ahn HJ, Kwon S, On YK, Lee JH, Cho Y, Oh IY, Lim HE, Cho MS, Nam GB, Lip GYH, Oh S. Reduction of AF Burden After Cryoballoon Ablation in Patients With Early Persistent AF: The COOL-PER Trial. JACC Clin Electrophysiol. 2025 Jun;11(6):1234-1247. doi: 10.1016/j.jacep.2025.02.006. Epub 2025 Mar 26. PMID 40146092